CLINICAL TRIAL: NCT02702635
Title: Measuring Blood Flow Characteristics Using Dynamic Contrast Enhanced Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5150234
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Brain Injuries; Cerebrovascular Disorders
MeSH Terms: conditions — Brain Injuries; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects (Experimental): All recruited subjects
  Interventions: Procedure: DCE MRI of the brain

INTERVENTIONS:
Procedure: DCE MRI of the brain — An MRI of the brain including a DCE sequence

SUMMARY:
Dynamic contrast-enhanced (DCE) MRI gives quantitative and semi-quantitative information about the integrity of the vascular system and can be used to quantify blood-brain barrier (BBB) integrity. The BBB plays a pathophysiological role in diabetes, cognitive disorders such as mild cognitive impairment, Alzheimer's disease, multiple sclerosis, and chronic traumatic encephalopathy. Although dysfunctional, changes in BBB integrity for these conditions are thought to be subtle and close to intact values. Recent studies have shown it is possible measure small changes in the BBB integrity as an early sign of disease using DCE MRI. The objective of this study is to apply an optimized DCE imaging protocol and novel image post-processing to obtain new information about the BBB integrity in aging. These techniques show promise for both improving clinical diagnosis, and elucidated the physiology or various disease processes.

DETAILED DESCRIPTION:
Objectives The objective of this investigator-initiated study is to continue and extend this research by applying our optimized DCE imaging protocol (using the standard FDA approved DCE sequence) and our novel image post-processing to obtain new information about the BBB integrity in aging.

Study Procedure Overview: Subjects will be recruited either from patient's at LLUMC with an existing order for a MRI study of the head with contrast, or from an exisiting cohort at LLU that participated in a previous study.

Health controls will be asked if they would like to participate in the study in order to evaluate if the optimized DCE sequence can provide useful information about various CNS diseases.

Imaging: Following consent, subjects will be imaged at LLUMC using the 3T MRI scanner (Siemens Medical Solutions, Malvern, PA) after MRI safety screening questionnaire is complete. Subjects will be asked to lie on or be positioned on their backs in the MRI scanner. The coil will be placed around their head and the subject will be provided with headphones and/or earplugs during the scan. Imaging will consist of the diagnostic MR protocol requested by the ordering physician and the addition of the standard FDA approved DCE sequence.

Data Collection and Analysis The collected DCE data may be processed using standard FDA approved DCE software (which the department already owns and uses clinically), used for clinical decision making purposes, and added to the patients record. The data will also be processed using specialized research software, this processing will not be used for diagnostic or clinical decision making purposes, and will not be added to the patients record. Ktrans values will be measured using region of interest analysis from the processed DCE data to determine if there are differences between the pathology of interest and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Any person between the ages of 0-100 years, who is undergoing routine magnetic resonance imaging (MRI) with contrast at LLUMC.

Or

• Any person between the ages of 18-100 years, who agrees to undergo routine magnetic resonance imaging (MRI) with contrast at LLUMC.

Exclusion Criteria:

* Electronic or metal implant that is not MRI safe, pregnancy or claustrophobia
* Not eligible for contrast agent injection (reduced renal function, GFR < 30 mL/min)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Correlation between Ktrans values and Omega3 levels | 2 years
Correlation between Ktrans values and neurocognitive testing | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Barnes, PhD, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No